CLINICAL TRIAL: NCT00510783
Title: IV Keppra in the Emergency Department for Prevention of Early Recurrent Seizures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Principal Investigator, Debra Houry, MD, MPH, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00002266; NCT00832858 (obsolete NCT alias)
Record Dates: First submitted 2007-07-31; First posted 2007-08-02 (Estimated); Results first posted 2013-08-05 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-11

CONDITIONS: Tonic-clonic Seizure
Keywords: tonic-clonic seizure; emergency department; IV levetiracetam; Keppra; seizures; phenytoin; Dilantin; Grand Mal seizure
MeSH Terms: conditions — Seizures; Emergencies; Epilepsy, Tonic-Clonic | interventions — Levetiracetam; fosphenytoin; Phenytoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phenytoin/Fosphenytoin (Active Comparator): Patients in the control arm will receive either IV Dilantin (1 gram of IV phenytoin infused at 25 mg/min or slower depending on vitals) or IV Fosphenytoin (1 gram of IV Fosphenytoin infused at 15 mg/min or slower depending on vitals).
  Interventions: Drug: Fosphenytoin; Drug: Dilantin
- Levetiracetam (Active Comparator): Patients in the intervention arm will receive IV Keppra (1 gram of Keppra added to 100 mL diluent infused over 15 minutes).
  Interventions: Drug: Keppra

INTERVENTIONS:
Drug: Keppra — The patient will receive 1 gram of Keppra added to 100ml diluent and will be infused over 15 minutes.
  Other Names: levetiracetam
  Arms: Levetiracetam
Drug: Fosphenytoin — IV load will be dependant on dilantin level. If no dilantin is detected in the patient, the patient will receive 1 gram of IV Fosphenytoin infused at 15 mg/min or slower depending on vitals.
  Other Names: Cerebyx
  Arms: Phenytoin/Fosphenytoin
Drug: Dilantin — IV load will be dependant on dilantin level. If no dilantin is detected in the patient, the patient will receive 1 gram of IV phenytoin infused at 25 mg/min or slower depending on vitals.
  Other Names: phenytoin
  Arms: Phenytoin/Fosphenytoin

SUMMARY:
This study is looking at three seizure medicines. Patients with seizures are usually treated with phenytoin (Dilantin) or Fosphenytoin. These medicines can be given intravenously (IV)or by mouth. Another seizure medicine, levetiracetam (Keppra) can now be given this way also. This study will compare IV phenytoin (Dilantin) and IV fosphenytoin to levetiracetam (Keppra) in patients who have had a recent seizure. Only patients with a history of seizures can be involved. The patient must present to the emergency department within 4 hours of a seizure. The purpose of this study is to compare these three drugs, phenytoin (Dilantin), fosphenytoin, and levetiracetam (Keppra). The investigators are looking to see if these drugs can prevent another seizure in the next 24 hours. We are also looking for any possible side effects.

DETAILED DESCRIPTION:
More than one in every one hundred patients presenting to the emergency department for care do so for seizures. More than half of these patients will require medications, often intravenously (IV), while in the emergency department. For many years the standard treatment has been phenytoin. However, there are many known contraindications to the use of this drug. These include known hypersensitivity, cardiac arrhythmias, cardiac disease, impaired liver or kidney function, diabetes mellitus, older age, thyroid disease, pregnancy, and alcohol use. A recent review of patients with seizure disorder at Emory Crawford Long and Emory University hospitals suggested that a significant percentage of those who were taking phenytoin actually had one or more of these contraindications. Additionally, the IV form of phenytoin has known, severe adverse effects including cardiovascular collapse, life threatening cardiac arrhythmias, and severe hypotension. There is another form of Phenytoin, called Fosphenytoin, that while safer in some respects still has similar concerns associated with its administration.

Levetiracetam (Keppra) has been available as an oral drug in the United States since 2000 and has a well established safety record when used as an add-on drug for patients with partial onset seizures. A double-blinded randomized study has shown that levetiracetam is also effective for primary generalized seizures as well.

The IV form of levetiracetam has recently been approved by the FDA for use. The only known contraindications other than known hypersensitivity include impaired renal function, psychiatric disorder, older age, and pregnancy. IV levetiracetam is not known to cause any of the acute, catastrophic events seen occasionally with phenytoin.

The investigators would therefore like to compare IV phenytoin and fosphenytoin to IV levetiracetam in preventing early recurrent seizures. Patients with known seizure disorders would be randomly assigned to one of two groups and therefore receive either IV fosphenytoin or IV levetiracetam. After an observation period, seizure free patients would be discharged and 24 hour phone follow up conducted to assess for the effectiveness of these anti-seizure medications as well as for any adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* patient presenting to Grady Memorial Hospital's Emergency Department after having a tonic-clonic seizure (primary or secondarily generalized) within the last 4 hours

Cause of seizure for inclusion: reason for seizure is often undetermined at time of presentation to the Emergency Department. The most likely expected causes of a seizure are noncompliance to existing antiepileptic drug regimen, refractory epilepsy with breakthrough seizure, metabolic aberration, alcohol withdrawal, or unknown.

Exclusion Criteria:

* non-English speaking
* first time seizure
* seizures other than tonic-clonic seizure (primary or secondarily generalized)
* more than 3 seizures in 24 hours or status epilepticus, pregnant patients by history or by urine pregnancy testing, serious neurologic insult resulting in seizure but where seizure is not the primary reason for admission (e.g. traumatic brain injury with seizure or hemorrhagic stoke would be excluded)
* contraindication to IV levetiracetam
* received IV phenytoin within 24 hours
* known allergy to phenytoin
* previously enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Houry, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study completed
Pre-assignment Details: study completed
Period: Overall Study
Arm/Group | Phenytoin/Fosphenytoin | Levetiracetam
Started | 82 | 76
Completed | 51 | 47
Not Completed | 31 | 29
Not completed — Lost to Follow-up | 29 | 25
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phenytoin/Fosphenytoin | Levetiracetam | Total
Number analyzed (Participants) | 82 | 76 | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 80 | 73 | 153
  >=65 years | 2 | 3 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 51.80 (106.459) | 65.79 (154.721) | 58.53 (131.651)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 53 | 109
  Male | 26 | 23 | 49
Region of Enrollment [Number; unit: participants]
  United States | 82 | 76 | 158

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Recurrent Seizure After Treatment.
Description: Recurrent seizure is defined as a seizure within 24 hours of treatment in the Emergency Department.
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Phenytoin/Fosphenytoin | Levetiracetam
Number analyzed (Participants) | 82 | 76
participants | 2 | 3

ADVERSE EVENTS:
Arm/Group | Phenytoin/Fosphenytoin | Levetiracetam
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/76
Other Adverse Events (participants affected / at risk) | 40/82 | 19/76
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phenytoin/Fosphenytoin (N=82) | Levetiracetam (N=76)
Fatigue (Investigations) | 4 (4) | 7 (7)
Burning at the IV Site (Investigations) | 11 (15) | 5 (5)
Itching (Investigations) | 8 (8) | 0 (0)
Dizziness (Investigations) | 17 (17) | 7 (7)

LIMITATIONS AND CAVEATS:
Several patients were lost to follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No